CLINICAL TRIAL: NCT00521742
Title: A Randomized, Double-Blind, Comparator-Controlled Study of Pioglitazone HCl vs Glyburide in the Treatment of Patients With Type 2 (Non-Insulin-Dependent) Diabetes Mellitus and Mild Cardiac Disease (NYHA I)
Brief Title: Efficacy of Pioglitazone Compared to Glyburide in Treating Subjects With Type 2 Diabetes Mellitus and Mild Cardiac Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-00-TL-OPI-520; U1111-1114-1616 (Registry Identifier: WHO)
Record Dates: First submitted 2007-08-25; First posted 2007-08-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pioglitazone 15 mg to 45 mg QD (Experimental)
  Interventions: Drug: Pioglitazone
- Glyburide 2.5 mg to 15 mg, QD (Active Comparator)
  Interventions: Drug: Glyburide
- Pioglitazone 15 mg or 30 mg QD (Experimental)
  Interventions: Drug: Pioglitazone
- Glyburide 5 mg or 10 mg, QD (Active Comparator)
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg to 45 mg, tablets, orally, once daily and glyburide placebo-matching capsules, orally, once daily for up to 52 weeks.
  Other Names: Actos; AD4833
  Arms: Pioglitazone 15 mg to 45 mg QD
Drug: Glyburide — Glyburide 2.5 mg to 15 mg, capsules, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 52 weeks.
  Arms: Glyburide 2.5 mg to 15 mg, QD
Drug: Pioglitazone — Pioglitazone 15 mg or 30 mg, tablets, orally, once daily and glyburide placebo-matching capsules, orally once daily for up to 52 weeks.
  Other Names: Actos; AD4833
  Arms: Pioglitazone 15 mg or 30 mg QD
Drug: Glyburide — Glyburide 5 mg or 10 mg, capsules, orally, once daily and pioglitazone placebo-matching tablets, orally once daily for up to 52 weeks.
  Arms: Glyburide 5 mg or 10 mg, QD

SUMMARY:
The purpose of this study is to evaluate the cardiovascular effects of pioglitazone, once daily (QD), versus glyburide when administered to patients with type 2 diabetes mellitus and mild cardiac disease.

DETAILED DESCRIPTION:
Diabetes is a chronic disease involving multiple metabolic defects that include inadequate insulin activity and resultant hyperglycemia. Individuals' differing genetic predisposition, level of physical activity, and age all contribute to variations in the onset and severity of type 2 diabetes. However, progression of this disease typically follows a characteristic pattern that begins as a reduced sensitivity of hepatic and peripheral-tissues to circulating insulin (ie, insulin resistance). The body's decreasing ability to produce adequate insulin to overcome insulin resistance (ie, insulin deficiency due to beta-cell insufficiency) results in impaired glucose tolerance and ultimately overt diabetes. In the United States, an estimated 17 million people have diabetes, with type 2 diabetes occurring in approximately 90% to 95% of cases.

The goal of treating type 2 diabetes is to control blood glucose and thereby prevent long-term complications. Adequate glycemic control is paramount in attempting to avert chronic complications, including blindness, renal dysfunction and resultant dialysis or renal transplantation, neuropathy, and nontraumatic amputations. Intensive glucose management in the early stages of diabetes may help forestall complications.

Pioglitazone is a thiazolidinedione developed by Takeda Chemical Industries, Ltd. Glyburide, is an oral antidiabetic agent of the sulfonylurea class. The primary purpose of this study is to evaluate the cardiovascular effects of pioglitazone versus glyburide when administered to patients with type 2 diabetes mellitus and mild cardiac disease

Study participation is anticipated to be approximately 1 year and 2 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Diagnosed with type 2 diabetes mellitus.
* Naive to oral antidiabetic pharmacologic therapy, who were currently taking sulfonylurea monotherapy, who were currently taking sulfonylurea/metformin combination therapy, or who were currently taking metformin monotherapy.
* Mild cardiac disease New York Heart Association functional Class I.
* Participated in dietary counseling.
* Glycosylated hemoglobin greater than or equal to 7.5% and less than 12% at Screening if naïve to oral antidiabetic pharmacologic therapy or taking metformin monotherapy, or greater than or equal to 6.5% and less than 12% if currently taking sulfonylurea monotherapy or taking ulfonylurea/metformin combination therapy.
* Stable therapy for cardiovascular dysfunction, defined as no change in therapy for greater than or equal to 4 weeks prior to Randomization.

Exclusion Criteria:

* Within the past 30 days treated with rosiglitazone, pioglitazone, or troglitazone or those previously treated with rosiglitazone, pioglitazone, or troglitazone but discontinued from therapy because of lack of efficacy or clinical or laboratory signs of intolerance.
* Treated with a sulfonylurea but discontinued for lack of efficacy or clinical or laboratory intolerance.
* Currently taking insulin or on continuous insulin therapy for control of their diabetes
* Type 1 (insulin-dependent) diabetes mellitus or a history of ketoacidosis.
* Any other investigational drug during the 30 days prior to Visit 1 or who will receive such a drug during the time-frame of this study.
* History of chronic alcoholism or drug abuse during the 6 months prior to the study.
* New York Heart Association functional Class II, III, or IV cardiac disease at Screening, or previous history of Class III or IV.
* Any of the following:

  * myocardial infarction
  * coronary angioplasty or bypass graft
  * unstable angina pectoris
  * transient ischemic attacks
  * documented cerebrovascular accident. 9. Abdominal, thoracic, or vascular surgery during the 3 months prior to Visit 1.
* Planned surgical or catheterization intervention within 6 months following Visit 1.
* Awaiting cardiac transplantation.
* Intercurrent illness severe enough to require hospitalization during the 3 weeks prior to Visit 1.
* Body mass index greater than 48 kg/m2 as calculated by [weight (kg)/height (m)2].
* Anemia having hemoglobin less than 10.5 g per dL for men and 10.0 g per dL for women.
* Triglyceride level greater than 500 mg per dL.
* Clinical evidence of active liver disease or alanine transaminase levels greater than 2.5 times the upper limit of normal.
* Serum creatinine greater than 2.0 mg per dL for men and 1.8 mg per dL for women or urinalysis protein (albumin) excretion levels greater than 2 plus on Combistix or equivalent and on repeat 24-hour results with greater than 3 g macroproteinuria.
* Unstable coronary syndromes.
* Systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 90 mm Hg at Screening.
* Serious uncontrolled cardiac rhythm disturbances.
* Symptomatic orthostatic hypotension or systolic blood pressure less than 90 mm Hg.
* Severe, advanced peripheral vascular disease (limb-threatening ischemia) or claudication resulting in the inability to walk greater than 1 block or to climb 10 stairs without interruption.
* Lower extremity amputation that would prevent the patient from performing the exercise test.
* Any other serious disease or condition which might affect life-expectancy or make it difficult to successfully manage and follow the subjects according to the protocol.
* Unexplained clinically significant findings on chest x-ray.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Oral, injected, or inhaled corticosteroids of greater than 2 week duration, or the need for recurrent us of corticosteroids.
  * Prescription niacin
  * Anti-diabetic medications except metformin
  * Cardiovascular medications must remain stable for at least 4 weeks prior to Randomization
  * Non-steroidal anti-inflammatory drugs
  * Aspirin greater than 325 mg per day

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2001-03; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Change in the walking distance during a standardized 6-minute walk test. | Weeks 2, 16, 24, 40, and 52 or Final Visit

SECONDARY OUTCOMES:
Morbidity and Mortality Due to Cardiovascular Events. | At occurrence or Weeks 2, 4, 6, 8, 12, 16, 24, 32, 36, 40, 48, and 52 or Final Visit
Change in Cardiovascular Treatment Program. | At occurrence or Weeks 2, 4, 6, 8, 12, 16, 24, 32, 36, 40, 48, and 52 or Final Visit
Change from Baseline in 12-lead Electrocardiogram Parameter (Ventricular Heart Rate) | Weeks 24 and 52 or Final Visit
Change from Baseline in Electrocardiogram Parameter (Left Ventricular Mass) | Week 52 or Final Visit
Change from Baseline in Electrocardiogram Parameter (Left Ventricular Ejection Fraction) | Week 52 or Final Visit
Change from Baseline in Electrocardiogram Parameter (Cardiac Index) | Week 52 or Final Visit
Change from Baseline in Electrocardiogram Parameter (Fractional Shortening) | Week 52 or Final Visit
Change in Blood Pressure | Weeks 2, 4, 6, 8, 12, 16, 24, 32, 40, 48, and 52 or Final Visit
Change in Heart Rate | Weeks 24 and 52 or Final Visit
Change in Body Weight | Weeks 2, 4, 6, 8, 12, 16, 24, 32, 40, 48, and 52 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda Global Research and Developmnet Center Inc

REFERENCES:
- [Result] Giles TD, Elkayam U, Bhattacharya M, Perez A, Miller AB. Comparison of pioglitazone vs glyburide in early heart failure: insights from a randomized controlled study of patients with type 2 diabetes and mild cardiac disease. Congest Heart Fail. 2010 May-Jun;16(3):111-7. doi: 10.1111/j.1751-7133.2010.00154.x. PMID 20557330
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI